CLINICAL TRIAL: NCT06924294
Title: Pattern and Short Term Outcomes of Renal Affection in Patients With Liver Cirrhosis in Al-Rajhi Liver Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Radwan Riad, Lecturer, Assiut University
Other Study IDs: liver cirrhosis
Record Dates: First submitted 2025-03-24; First posted 2025-04-11 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Liver Cirrhosis
Keywords: renal affection in patients with liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- liver cirrhosis admitted to Al-Rajhi liver hospital: observation of renal affection in patients known to have liver cirrhosis
  Interventions: Other: observation of renal affection in patients with liver cirrhosis

INTERVENTIONS:
Other: observation of renal affection in patients with liver cirrhosis — * CBC
  * Liver function test
  * kidney function test (serum creatinine, BUN, eGFR (EPI equation and MDRD equation) ,
  * Prothrombin time and concentration, INR,
  * Serum electrolytes
  * Urine analysis.

SUMMARY:
* To characterize the pattern and the prevalence of renal affection among liver cirrhosis patients.
* To evaluate the short-term outcomes of those patients.

DETAILED DESCRIPTION:
Liver cirrhosis is a chronic liver disease characterized by significant scarring and dysfunction. One of its common complications is renal affection , which can significantly impact patient outcomes .

Aetiology of AKI can be categorized into three main types. These are prerenal (results from decreased renal perfusion), intrinsic renal (acute tubular necrosis), and postrenal AKI. In patients on admission, acute tubular necrosis is a common type of intrinsic AKI .

The development of portal hypertension in patients with liver cirrhosis leading to a reduction in systemic vascular resistance as a result of primary arterial vasodilation in the splanchnic circulation is the primary cause of AKI in cirrhotics. This mechanism primarily leads to hepatorenal syndrome. In addition, the underlying causes of liver cirrhosis can be the cause of intrinsic renal disease .

Early identification and management of AKI may improve outcomes. AKI in patients with liver cirrhosis in Egypt and their impact on inpatient mortality are largely unknown. This study was aimed at determining the prevalence, precipitating factors, predictors, and in-hospital mortality of AKI in patients with liver cirrhosis admitted at Al-Rajhi liver hospital at Egypt .

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis admitted to the department .

Exclusion Criteria:

1. Patients with known preexisting chronic kidney disease according to KDIGO and EASL 2018 definitions ( defined as functional GFR <60 ml/min per 1.73 m 2 for ≥3 months or structural kidney damage for ≥3 months ).
2. Patient refusal to give informed consent ( or his first degree relatives in case of disturbed conscious level).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with liver cirrhosis admitted to the department .
Sampling Method: Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | Through the study completion , average 6 months
  Mortality during hospital stay
Phenotypes of acute kidney injury across geographic areas | Baseline ( at admission ), then through the study completion, average 6 months
  Characteristics of acute kidney injury (clinical type and stage)

SECONDARY OUTCOMES:
28-day mortality | 28 days
  Mortality at 28 days
Resolution of AKI | Hospital stay (up to 90 days)
  Resolution of AKI will be defined as return of serum creatinine to a value within 0.3 mg/di (26.5 mmol/L) of the baseline value. Partial response will be defined as regression of AKI to a lower stage with a reduction of serum creatinine to ≥0.3 mg/d| (26.5 mmol/L) above the baseline value
Development of CKD | 90 days
  Chronic kidney disease will be defined as an estimated glomerular filtration rate <60 ml/min ml/min/1.73 m2 for >3 months. The Modification of Diet in Renal Disease equation will be used for estimating glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Omar Abd El-Malek, professor, Study Director — Assiut University
Locations (1):
- Al-Raghi liver hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi YJ, Kim JH, Koo JK, Lee CI, Lee JY, Yang JH, Ko SY, Choe WH, Kwon SY, Lee CH. Prevalence of renal dysfunction in patients with cirrhosis according to ADQI-IAC working party proposal. Clin Mol Hepatol. 2014 Jun;20(2):185-91. doi: 10.3350/cmh.2014.20.2.185. Epub 2014 Jun 30. PMID 25032185
- [Background] Duah A, Nkrumah KN. Prevalence and predictors for spontaneous bacterial peritonitis in cirrhotic patients with ascites admitted at medical block in Korle-Bu Teaching Hospital, Ghana. Pan Afr Med J. 2019 May 16;33:35. doi: 10.11604/pamj.2019.33.35.18029. eCollection 2019. PMID 31384350
- See also: https://scholar.google.com/scholar_lookup?journal=Clinical%20and%20Molecular%20Hepatology&title=Prevalence%20of%20renal%20dysfunction%20in%20patients%20with%20cirrhosis%20according%20to%20ADQI-IAC%20working%20party%20proposal&author=Y.%20J.%20Choi&author — https://GoogleScholar.com